CLINICAL TRIAL: NCT05708586
Title: Virtual Reality Decreases Child Anxiety and Pain as Well as Caregiver Anxiety and Pain Perception During Orthopaedic Clinic Office Procedures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary findings showed no significant difference between virtual reality and distraction techniques.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Noelle Whyte, Clinical Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00197192
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Anxiety; Pain
Keywords: Virtual reality
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (Active Comparator): Standard comfort given
  Interventions: Behavioral: Control
- Virtual Reality (VR) (Experimental)
  Interventions: Device: Virtual Reality (VR)

INTERVENTIONS:
Behavioral: Control — This is the control condition and anxiety is addressed in a standard way of having the care taker calm the child during the intervention.
  Arms: Control
Device: Virtual Reality (VR) — The child who is undergoing a procedure uses VR as a distraction during the intervention
  Arms: Virtual Reality (VR)

SUMMARY:
The purpose of this study is to demonstrate that the use of a virtual reality experience can decrease child and caregiver anxiety and pain for simple orthopaedic office procedures.

ELIGIBILITY:
Inclusion Criteria for pediatric patient:

* Undergoing cast removal, pin removal, or suture removal in study affiliated clinic
* Less than 17 years old

Exclusion Criteria for pediatric patient:

* History of seizures
* Pregnant, have preexisting binocular vision abnormalities or psychiatric disorders, or suffer from a heart condition or other serious medical condition
* Patients can't have implanted medical devices including cardiac pacemakers, hearing aids and defibrillators

There is no minimum or maximum age for the Caretakers/Parents.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Whyte, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 66 participants listed in the registration, three participants' data became unusable during the study, and therefore cannot be a part of the record. Parents of the children enrolled were asked to respond to a survey on a voluntary basis, but were not enrolled in the study as participants, did not contribute baseline data, and were not required to respond to the survey as part of their child's participation.
Period: Overall Study
Arm/Group | Control | Virtual Reality (VR)
Started | 28 | 35
Completed | 28 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Virtual Reality (VR) | Total
Number analyzed (Participants) | 28 | 35 | 63
Age, Customized [Count of Participants; unit: Participants]
  Age <7 | 8 | 7 | 15
  Age >=7 | 20 | 28 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 14 | 19 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28 | 35 | 63

OUTCOME MEASURES:

1. Primary Outcome: Child Pain Score
Description: Assessed by Wong-Baker Children's Faces Pain Scale: The scale shows a series of faces ranging from a happy face at 0 which represents "no hurt" to a crying face at 10 which represents "hurts worst." Based on the faces and descriptions, the patient chooses the face that best describes their level of pain.
Time Frame: Up to 24 hours following procedure
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | Virtual Reality (VR)
Number analyzed (Participants) | 28 | 35
units on a scale
  Pre-Intervention | .5 [0 to 6] | 1.2 [0 to 4]
  Post-Intervention | 1.07 [0 to 10] | .97 [0 to 6]

2. Primary Outcome: Child Anxiety (7 Years Old and Older)
Description: Assessed by State-Trait Anxiety Inventory for Children (STAIC): 20 questions with 3 answer options for each question.
  Scores range from 20 to 60 with 60 being the higher (more or worse) anxiety on self-assessment.
Time Frame: Up to 24 hours following procedure
Population: Note: This data is only for participants 7 and older, as also shown in baseline characteristics.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | Virtual Reality (VR)
Number analyzed (Participants) | 20 | 28
units on a scale
  Pre-Intervention | 28.55 [20 to 42] | 32.88 [20 to 46]
  Post-Intervention | 26.35 [20 to 31] | 27.96 [20 to 47]

3. Primary Outcome: Child Anxiety (Younger Than 7 Years Old)
Description: Assessed by Children's Fear Scale: The Children's Fear Scale (CFS) is used to measure the anxiety or fear level of the children. The one-item scale consists of a row of five sex neutral faces ranging from a no fear (neutral) face on the far left to a face showing extreme fear on the far right. Thus, the scale is 1-5 with 1 being least fear and 5 being greatest fear and anxiety.
Time Frame: Up to 24 hours following procedure
Population: Note: This data is only for participants younger than 7 years old, as also shown in baseline characteristics.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | Virtual Reality (VR)
Number analyzed (Participants) | 8 | 7
units on a scale
  Pre-Intervention | 1.375 [0 to 4] | 1.5 [0 to 4]
  Post-Intervention | .75 [0 to 4] | 0.875 [0 to 4]

4. Secondary Outcome: Parental Anxiety
Description: Assessed by State-Trait Anxiety Inventory (STAI): a 20 question inventory where each question is on a Likert scale 1-4. The total range of the inventory is 20-80 with higher scores indicating more anxiety (please note that some questions are reverse coded).
Time Frame: Up to 24 hours following procedure
Population: Data was volunteered by 63 parents or caretakers of the participants. They were not consented separately from the children who were the focus of the study.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Control | Virtual Reality (VR)
Number analyzed (Participants) | 28 | 35
score on a scale | 46.61 [34 to 65] | 46.91 [37 to 61]

ADVERSE EVENTS:
Time Frame: Up to 24 hours
Arm/Group | Control | Virtual Reality (VR)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/35
Other Adverse Events (participants affected / at risk) | 0/28 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT05708586/Prot_000.pdf